CLINICAL TRIAL: NCT03943719
Title: The Impact of a Rapid Molecular Identification Test on Positive Blood Cultures From Critically Ill With Bacteremia: a Pre-post Intervention Study
Brief Title: Clinical Impact of the FilmArray Blood Culture Identification Panel Performed on Positive Blood Cultures From Intensive Care Patients With Septicemia
Acronym: SEPSIS2016
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: SEPSIS2016; 2016/19SEP/401 (Other: CEHF)
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Septicemia
Keywords: FilmArray; bacteremia; septicemia; clinical impact; molecular testing; identification; positive blood culture; optimal antimicrobial treatment
MeSH Terms: conditions — Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FilmArray blood culture identification panel — FilmArray blood culture identification panel is performed 24 hours on 24hours and 7 days a week on positive blood cultures to accelerate pathogens detection

SUMMARY:
Molecular testing is a largely validated approach allowing rapid identification of positive blood cultures. However, due to its high cost and its limited information on susceptibility, it is considered as an add-on technique reserved for specific patient populations. In our study, we specifically evaluated molecular testing in a critical care setting and measured its impact on the therapeutic management of critically ill with positive blood cultures. Through the analysis of 110 positive blood culture episodes included in both pre- and post intervention period, we measured a drastic 14h-reduction of the time to administration of the optimal antimicrobial treatment with the use of the molecular approach.

ELIGIBILITY:
Inclusion Criteria:

* adult intensive care unit patients with positive blood cultures

Exclusion Criteria:

* palliative care patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult intensive care unit patients with positive blood cultures
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Turn Around Time to optimal treatment of septicemia | From positivity detection of positive blood culture to administration of optimal treatment (up to 48 hours)
  Time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alexia VERROKEN, Principal Investigator — Cliniques universitaires St-Luc
Locations (1):
- Cliniques universitaires St-Luc, Brussels, Belgium